CLINICAL TRIAL: NCT02575612
Title: Can a Pathological Complete Response in the Breast be Diagnosed by Vacuum-assisted, Ultrasound Guided Minimal Invasive Biopsy After Neoadjuvant Chemotherapy in Breast Cancer Patients? A Proof of Concept From a Prospective Cohort Study
Brief Title: Diagnosis of Pathological Complete Response by Minimal Invasive Biopsy After Neoadjuvant Chemotherapy in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Jörg Heil, Prof. Dr. med Jörg Heil, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vacuum-assisted biopy (Experimental): All patients enrolled in this study received a vacuum-assisted biopsy before surgery.
  Interventions: Procedure: vacuum-assisted biopsy

INTERVENTIONS:
Procedure: vacuum-assisted biopsy — Ultrasound guided VAB was used directly prior to breast conserving surgery or mastectomy. It was performed by experienced physicians (> 50 ultrasound guided minimal invasive biopsies per year, > 500 breast ultrasound examination of the breast per year). The needle was placed below or beside the target lesion according to physician's choice. At least six biopsies should be taken; up to 12 according to the physicians choice. After the VAB a clip marker was placed to highlight the position of the biopsy for specimen radiography and pathology.
  Other Names: VAB; vacuum-assisted minimal invasive biopsy

SUMMARY:
The study aims to evaluate the ability of representative vacuum-assisted minimal invasive biopsy (VAB) to diagnose pathological complete response (pCR=ypT0) in breast cancer patients after neoadjuvant chemotherapy (NACT).

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NACT) is an increasingly used approach for patients with locally advanced and primarily inoperable breast cancer or for patients with potentially chemosensitive tumors. In clinical routine surgical treatment follows the pre-operative chemotherapy. However, recent studies have demonstrated that shrinking tumors need less surgical treatment indicating that patients with pCR could potentially be spared of surgery in the future.

Up to now, prediction of pCR after NACT, i.e. diagnosing a pCR without surgery, is based on tumor biology at diagnosis, the applied NACT regimen and breast imaging results; all with mediocre accuracy. This prospective, monocenter diagnostic trial aims to explore if minimal invasive biopsies (MIB) might overcome this diagnostic challenge.

From September 1st, 2014 to February 15th, 2015 the investigators performed ultrasound guided vacuum-assisted minimal invasive biopsy (VAB) on 50 breast cancer patients after NACT and directly prior to surgery. To analyse VAB pathologically results were categorized as follows: residual vital tumor cells (invasive, in situ, both, lymphangiosis carcinomatosous) present, (significant parts of) the tumor bed present, neither vital tumor cells nor (significant parts of) the tumor bed (indicating a non representative VAB). The results were compared to those of the pathological examination of surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

The investigators included patients

* after neoadjuvant chemotherapy (NACT) according to the NACT protocol
* with at least one detectable mass / marker after NACT in ultrasound
* with cT1c-cT4a-c tumors
* after informed consent
* with unilateral or bilateral primary breast cancer, confirmed histologically prior to chemotherapy
* with known grading, ER/PgR/HER-2neu- and Ki-67 status
* with breast ultrasound, mammography (and breast MRI where necessary) before and after NACT
* clinical / imaging partial or complete response to NACT

Exclusion Criteria:

The investigators excluded patients from the study with

* NACT <12 weeks because of termination due to progressive disease, massive adverse events or patient wish
* non-detectable mass in ultrasound / dislocation of marker (> 10mm distance to the initial lesion)
* cT4d stage (inflammatory breast cancer)
* M1 stages
* stable disease according to a multimodal assessment of ultrasound, mammography and breast MRI (if available) according to RECIST

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
false negative rate to diagnose a pathological complete response by vacuum-assisted biopsy for the whole cohort and predefined subgroups | 1 week
  As an explorative study, the statistical analysis was performed using descriptive methods only.
  For a baseline comparison between groups, the investigators compared the group of patients with pCR to the group of patients without pCR. As primary outcomes the investigators calculated negative predictive values (NPV) and false negative rates (FNR) for the whole study cohort as well as for certain subgroups (especially addressing the question of evaluating representativeness of VAB). The investigators calculated two-sided-95% confidence intervals for all results.

SECONDARY OUTCOMES:
negative predictive values to diagnose a pathological complete response by vacuum-assisted biopsy for the whole cohort and predefined subgroups | 1 week
  As an explorative study, the statistical analysis was performed using descriptive methods only.
  For a baseline comparison between groups, the investigators compared the group of patients with pCR to the group of patients without pCR. As primary outcomes the investigators calculated negative predictive values (NPV) and false negative rates (FNR) for the whole study cohort as well as for certain subgroups (especially addressing the question of evaluating representativeness of VAB). The investigators calculated two-sided-95% confidence intervals for all results.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Heil, Prof. Dr., Study Chair — University of Heidelberg, Department of Gynecology, Breast Unit
Locations (1):
- University Breast Unit, Department of Gynecology, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Pfob A, Sidey-Gibbons C, Rauch G, Thomas B, Schaefgen B, Kuemmel S, Reimer T, Hahn M, Thill M, Blohmer JU, Hackmann J, Malter W, Bekes I, Friedrichs K, Wojcinski S, Joos S, Paepke S, Degenhardt T, Rom J, Rody A, van Mackelenbergh M, Banys-Paluchowski M, Grosse R, Reinisch M, Karsten M, Golatta M, Heil J. Intelligent Vacuum-Assisted Biopsy to Identify Breast Cancer Patients With Pathologic Complete Response (ypT0 and ypN0) After Neoadjuvant Systemic Treatment for Omission of Breast and Axillary Surgery. J Clin Oncol. 2022 Jun 10;40(17):1903-1915. doi: 10.1200/JCO.21.02439. Epub 2022 Feb 2. PMID 35108029
- [Derived] Pfob A, Sidey-Gibbons C, Lee HB, Tasoulis MK, Koelbel V, Golatta M, Rauch GM, Smith BD, Valero V, Han W, MacNeill F, Weber WP, Rauch G, Kuerer HM, Heil J. Identification of breast cancer patients with pathologic complete response in the breast after neoadjuvant systemic treatment by an intelligent vacuum-assisted biopsy. Eur J Cancer. 2021 Jan;143:134-146. doi: 10.1016/j.ejca.2020.11.006. Epub 2020 Dec 8. PMID 33307491